CLINICAL TRIAL: NCT01632111
Title: Impact of the Treatment With Agalsidase Alpha on Lung Function and on Pulmonary Involvement in Patients With Fabry Disease. A Multicenter, Retrospective Observational Study
Brief Title: Pulmonary Involvement in Patients With Fabry Disease
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Fabry
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — Vital Capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Lung function measurement — Spirometry
  Other Names: FEV1, FVC

SUMMARY:
The objective of this study is to investigate whether Agalsidase alpha, a drug commonly prescribed in patients with Fabry disease, is associated with improvement of the pulmonary involvement. According to the Global Initiative for Obstructive Lung Disease (GOLD), the surrogate markers for obstructive lung diseases are a decrease in both forced expiratory volume in one second (FEV1) and FEV1/FVC ratio, whereas FVC is the forced vital capacity. However, the measurement of these lung function parameters is indicated as yearly follow-up examinations with or without the treatment of Agalsidase alpha in patients with Fabry disease.

DETAILED DESCRIPTION:
Pulmonary function tests und DLCO measurements are performed yearly in relation with yearly follow up examinations in the Department of Internal Medicine from the University Hospital of Zurich. We will retrospectively collect the results of the pulmonary functions test (spirometry).

ELIGIBILITY:
Inclusion criteria:

* All patients with established diagnosis of Fabry disease

Exclusion criteria:

* Missing informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ambulatory patients at University Hospital of Zurich with Fabry disease
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Lung function measurements | From first consultation until present
  Retrospective analysis of yearly measured lung function parameters to investigate on the lung function changes in patients with Fabry disease

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — University Hospital Zurich, Division of Internal Medicine
Locations (1):
- University Hospital Zurich, Division of Internal Medicine, Zurich, Switzerland